CLINICAL TRIAL: NCT06925958
Title: A Clinical Trial Evaluating the Safety Tolerability, Radiation Absorption Dose, Distribution, PET Imaging and Histological Expression of 68Ga-NOTA-SCH001 in Patients With Multiple Myeloma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-MI- 68Ga-NOTA-SCH001-34
Record Dates: First submitted 2025-03-27; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma (MM)
MeSH Terms: conditions — Multiple Myeloma | interventions — Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-NOTA-SCH001 PET/CT imaging (Experimental)
  Interventions: Diagnostic Test: Flow cytometry

INTERVENTIONS:
Diagnostic Test: Flow cytometry — CD38 Flow cytometry testing

SUMMARY:
Multiple myeloma is the second most common hematologic malignancy in adults, and no curative treatment currently exists. With the development of monoclonal antibodies for tumor therapy, identifying tumor-specific biomarkers has become a prerequisite for pre- and post-treatment evaluation. CD38, which is abnormally elevated in 95% to 100% of malignant plasma cells but relatively low in normal cells, serves as a biomarker for multiple myeloma. In clinical practice, CD38 expression is typically detected through flow cytometry and microscopic examination of bone marrow biopsy samples. However, biopsies are invasive and prone to false-negative results in cases of heterogeneity or small lesion samples, whereas whole-body imaging methods allow non-invasive assessment of target expression.

[¹⁸F]FDG PET/CT imaging is one of the most commonly used techniques in multiple myeloma. However, its diagnostic application is limited by false-negative results due to low hexokinase 2 expression in myeloma cells. Additionally, it fails to provide accurate molecular information, such as CD38 expression in cells. Therefore, this study aims to develop a more specific and stable molecular imaging probe, ⁶⁸Ga-NOTA-SCH001, to non-invasively visualize CD38 expression and monitor responses to CD38-targeted therapy in real time. This approach may also contribute to the formulation and optimization of clinical treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* 1. The subjects sign the informed consent voluntarily and can complete the test according to the protocol requirements;

  2. Over 18 years old, male or female;

  3. Patients diagnosed with multiple myeloma;

  4. ECOG score is 0-1; The expected survival time is not less than 3 months;

  5. Women of childbearing age need to undergo urine pregnancy test, and enrolled patients must be negative for pregnancy test;

  6. For fertile female patients or male patients with fertile partners, agree to remain abstinent during the study period (no

Or use one or more contraceptive methods with a failure rate of less than 1% per year for at least one year after the end of the study.

7. CD38 monoclonal antibody therapy was not used before enrollment in this study.

Exclusion Criteria:

* General situation

  * Those who are unable to perform visits, or receive relevant tests, or treatment in accordance with the clinical trial protocol;
  * Can not tolerate venous puncture blood collection;
  * Patients with serious diseases or other malignant tumors, except those that the researchers determined to be in stable control;
  * Known severe allergy to SCH001, similar drugs or excipients;

Laboratory examination

• Serum virology test: any of the results of hepatitis B virus surface antigen, hepatitis C virus antibodies, syphilis specific antibodies

Positive or HIV-negative antibodies cannot be determined;

• Fasting blood glucose >11.1mmol/L;

other

* No active infection
* Drug/alcohol abuse, severe mental disorders;
* Patients with claustrophobia, emotional instability, acute persistent spasms, or inability to keep their arms up and lie flat for 30 minutes;

Participants in any other clinical trial within 3 months prior to screening;

* Women who are pregnant or breastfeeding;
* The investigator did not consider it appropriate to participate in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
PET/CT imaging SUV value | 0-30minutes、60minutes、120minutes